CLINICAL TRIAL: NCT07350603
Title: Using Inclusive Art Participation as a Means to Promote Psychosocial Health Among People With Physical Disabilities in Residential Care Homes: A Mixed-Methods Feasibility Study
Brief Title: Using Art Participation to Promote Psychosocial Health Among People With Physical Disabilities: A Feasibility Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Nethersole School of Nursing (Other)
Responsible Party: Principal Investigator, Mimi Wai Man Chan, Dr., The Nethersole School of Nursing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22385
Record Dates: First submitted 2025-12-31; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Physical Disability
Keywords: Art; Residential care home; Feasibility; Mixed-methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Art intervention (Experimental)
  Interventions: Other: Inclusive art program

INTERVENTIONS:
Other: Inclusive art program — The inclusive art participation program will consist of a six-weekly session syllabus of 90 minutes per session. It will be led by a nurse facilitator who has been trained in using art as a healing tool in the healthcare context. Group format of four to six participants per group will be adopted. It will be conducted in a private and active room at residential care homes, which offers a comfortable space that enables participants to express themselves in a safe and confidential environment. The program will focus not only on promoting psychosocial health but also emphasize the inclusive and supportive environment to contribute to social interaction and engagement in meaningful social activities, that affirm the rights of people with physical disabilities living in residential settings.

SUMMARY:
This study aims to explore the feasibility of a newly developed theory-based inclusive art participation program for promoting psychosocial health of people with physical disabilities living in residential care homes.

Specifically, the feasibility is assessed following the framework proposed by Bowen et al. (2009), which encompassed five aspects, including demand, implementation, practicality, preliminary effects, and acceptability. As for the preliminary effects, this project will evaluate self-esteem, sense of control, self-efficacy, mood, and social connectedness after the completion of program.

This study will adopt a one group pretest-posttest approach with quasi-experimental design to collect both quantitative and qualitative data, employing a mixed-methods study design.

DETAILED DESCRIPTION:
The World Health Organization (WHO) estimates that approximately 1.3 billion people, around 16% of the global population, are currently living with disabilities, encompassing mental, intellectual, and physical disabilities. Among those, over 30% of them experience physical disabilities. These numbers reflect that a large proportion of people in global experience mobility, dexterity, coordination, or stamina impairments, which may result from traumatic injuries, nervous system disorders, autoimmune diseases, or age related degenerative diseases. As a result, some people with physical disabilities are unable to take care of themselves and thus require assistance from family members or caregivers, while some further consequently reside in residential care homes to receive ongoing support.

Although residential care homes offer essential medical and daily living support to people with physical disabilities who cannot be taken care of at home, these facilities have mainly prioritized physical care. While psychosocial needs are often addressed as a secondary concern or sometimes overlooked. On the other hand, current evidence reports that some residents with physical disabilities spend much of time physically and socially inactive. Due to limitation in mobility, many of them may not independently perform basic activities of daily living or engage in social interactions, which may bring a great loss of autonomy, competence, and relatedness to them, leading to psychosocial health issues.

In recent decades, there has been an increasing interest in the use of art participation in healthcare settings to serve as a multidisciplinary approach to facilitate health of individuals. Growing evidence also supports the positive impact of art participation on psychosocial health of individuals in residential settings. Nevertheless, such evidence focuses on the population of older adults, people with dementia, and children with intellectual disabilities, while the benefits of people with physical disabilities in residential settings remain unclear. Furthermore, the scope of such evidence primarily underscores art participation as a tool for addressing health issues by non-verbal expression and non-judgmental environments. However, it overlooks the potential of art participation as a valued and inclusive social activity that affirms the rights of people with physical disabilities, meanwhile, contributes meaningfully to their psychosocial health. Moreover, there is a lack of understanding of the processes by which art participation supports communication, expression, choice, and autonomy of people with physical disabilities. Clearly, pediatric inclusive art participation program within residential settings requires both evidence and theory to move forward as a recognized program format. Based on such evidence, there is a need to conduct a more specific study that focuses on using inclusive art participation programs for residents with physical disabilities who experience physical and social barriers.

Due to the lack of research on the continued examination of how the process of inclusive art participation benefit people with physical disabilities in residential care homes, developing a new inclusive art participation program for them is warranted to investigate its impacts. More importantly, the Medical Research Council (MRC) framework suggests that the stage of feasibility should be conducted to assess the procedure for developing and evaluating a complex program and to determine whether the definitive study can be undertaken in the future. Therefore, it is worthwhile designing a study to explore the feasibility of this newly developed program prior to conducting a large-scale study to examine its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years old or above
* have single or multiple physical disabilities caused by disease, accident, or aging, characterized by long-term impairments in mobility, stamina, or dexterity
* reside in residential care home
* only have a mild cognitive impairment defined as having a Montreal Cognitive Assessment (MoCA) score which fall above the 16th percentile
* have upper limb function with below a score of 50 assessed by Quick Disability of the Arm, Shoulder and Hand (DASH) Questionnaire
* able to remain in sitting position independently
* able to understand and communicate with Chinese, and (8) able to read Traditional Chinese.

Exclusion Criteria:

* individuals with severely impaired speaking, hearing, or visual acuity
* individuals have physical unwell for participating in this study
* individuals are currently taking part in other research projects or receiving other programs for promoting psychosocial health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Preliminary effects - Sense of control | From enrollment to the end of treatment at 6 weeks.
  The Chinese version of Recovery Locus of Control Scale (RLOCS) 9-item will be adopted to assess sense of control. Each item is rated on a five-point scale from 1='strongly agree' to 5='strongly disagree'. The total score ranged from 9 to 45. A higher total score indicates a better sense of control.
Preliminary effects - Self-esteem | From enrollment to the end of treatment at 6 weeks.
  The Chinese version of Rosenberg Self-Esteem Scale - 10-item (RSES) will be adopted to measure self-esteem. It consists of five positively worded items and five negatively worded items. Each item is rated on a four-point scale. Specifically, positively worded items are given a score from 1='strongly agree' to 4='strongly disagree', while negatively worded are reverse scored, from 1='strongly disagree' to 4='strongly agree'. The total score is summed up to give a range from 10 to 40. A higher score represents greater self-esteem.
Preliminary effects - Self-efficacy | From enrollment to the end of treatment at 6 weeks.
  The Chinese version of General Self-Efficacy Scale (GSES) 10-item will be used to measure self-efficacy. Each item is rated on a four-point scale from 1='not at all true' to 4='exactly true'.The total score is summed up to give a range from 10 to 40. A higher score represents greater general self-efficacy.
Preliminary effects - Mood | From enrollment to the end of treatment at 6 weeks.
  The Chinese version of Positive and Negative Affect Scale (PANAS) will be used to evaluate mood. It is a 20-item self-report questionnaire that measures mood by assessing the experience of positive and negative emotions, which are 10 items for positive emotions and other 10 items for negative emotions. Each item is rated on a five-point scale from 1=' very slightly or not at all' to 5='extremely'. The total scores range from 10 to 50 for positive and negative mood, respectively. A higher score of positive domain indicates higher levels of positive affect, while a lower score of negative domain represents lower levels of negative affect.
Preliminary effects - Social connectedness | From enrollment to the end of treatment at 6 weeks.
  The Chinese version of Social Connectedness Scale - Revised - 20-item (SCS-R) to assess social connectedness. Each item is rated on a six-point scale from 1='strongly disagree' to 6='strongly agree'. The total score is summed up to give a range from 20 to 120. A higher score indicates more connectedness to others.

OTHER OUTCOMES:
Demand | From enrollment to the end of treatment at 6 weeks.
  Demand in this study refers to recruitment rate. Recruitment rate will be calculated by the following formula: the numbers of participant recruited in the program over the total numbers of potential participant approached.
Practicality | From enrollment to the end of treatment at 6 weeks.
  Practicality in this study means adverse events. Adverse events will be narratively recorded in a team-developed observation note sheet.
Implementation | From enrollment to the end of treatment at 6 weeks.
  Implementation in this study refers to attrition rate. Attrition rate will be calculated by the following formula: the numbers of participant dropped out of the study over the numbers of participant recruited in this study.
Acceptability | After the end of treatment at 6 weeks.
  Acceptability in this study means participants' experiences and perspectives of engaging in the program. A team-developed interview guide will be adopted to collect such data.

IPD SHARING:
Plan to Share IPD: No